CLINICAL TRIAL: NCT05869565
Title: A Randomized, Blinded, Placebo-Controlled Phase 2B Clinical Trial to Compare the Efficacy of Different Combinations of Sodium Chloride and Sodium Acetate IV Fluids Along With Standard of Care Treatment in Acute Stroke Patients.
Brief Title: Best Solution Identification to Prevent Hyperchloremia Combinations of Sodium Chloride and Sodium Acetate IV Fluids Along With Standard of Care Treatment in Acute Stroke Patients
Acronym: sodium acetate
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Zeenat Qureshi Stroke Institute (Other)
Responsible Party: Principal Investigator, MUHAMMAD WASAY, professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-7608-22106
Record Dates: First submitted 2023-04-18; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: A Randomized, Blinded, Placebo-Controlled phase 2B clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Randomized, Blinded, Placebo-Controlled phase 2B clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Normal saline arm (Active Comparator): Sodium chloride (0.9%) referred as 0.9% NaCl for 72 hours post symptom onset (60-72 hourspost randomization);
  Interventions: Drug: Sodium Chloride 0.9% infusion alone or in combination with Sodim acetate with normal saline in a ratio 1;1, 2;1 and 3;1
- normal saline sodium acetate 3;1 (Active Comparator): Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 3:1 ratio for 72 hours post symptom onset (60-72 hours post randomization
  Interventions: Drug: Sodium Chloride 0.9% infusion alone or in combination with Sodim acetate with normal saline in a ratio 1;1, 2;1 and 3;1
- normal saline sodium acetate 2;1 (Active Comparator): Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 2:1 ratio for 72 hours post symptom onset (60-72 hours post randomization);
  Interventions: Drug: Sodium Chloride 0.9% infusion alone or in combination with Sodim acetate with normal saline in a ratio 1;1, 2;1 and 3;1
- normal saline sodium acetate 1;1 (Active Comparator): Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 1:1 ratio for 72 hours post symptom onset (60-72 hours post randomization).
  Interventions: Drug: Sodium Chloride 0.9% infusion alone or in combination with Sodim acetate with normal saline in a ratio 1;1, 2;1 and 3;1

INTERVENTIONS:
Drug: Sodium Chloride 0.9% infusion alone or in combination with Sodim acetate with normal saline in a ratio 1;1, 2;1 and 3;1 — Patients will be enrolled in the study and randomized into one of four arms
  Other Names: Sodim chloride alone; sodium chloride with sodium acetate ratio 3;1; sodium chloride with sodium acetate ratio 2;1; sodium chloride and sodium acetate ratio 1;1

SUMMARY:
Hypothesis:

Hyper chloremia is associated with poor outcome in Intracerebral Hemorrhage (ICT). Hyperchloremia is defined as serum chloride level of 110mmol/L or greater. This clinical study is assuming that, by increasing the ratio of Sodium-acetate to Sodium-chloride solutions in IV treatment, the incidence of Hyperchloremia can be lowered significantly. This result can be demonstrated by measuring serum chloride levels at Baseline, 24Hr, 48Hr and 72 Hours' time intervals and compare them between the three treatment and one Control arm.

Intervention (drug/biologic/device/behavioral):

Phase 2-dose finding Patients will be enrolled in the study and randomized into one of the four study treatment arms(target fluid administration rate 1 ml/kg/hour) initiated within 12 hours. IVF will be prepared in the main hospital pharmacy.

1. Sodium chloride (0.9%) referred as 0.9% NaCl for 72 hours post symptom onset (60-72 hourspost randomization);
2. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 3:1 ratio for 72 hours post symptom onset (60-72 hours post randomization);
3. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 2:1 ratio for 72 hours post symptom onset (60-72 hours post randomization);
4. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 1:1 ratio for 72 hours post symptom onset (60-72 hours post randomization).

DETAILED DESCRIPTION:
Background and Rational:

Acute stroke and intracerebral hemorrhages are most common admissions in neurological intensive care units. Proper management of these diseases helps to achieve better outcomes and reduce the burden on family and society. Proper volumes and concentration of intravenous fluids maintains sufficient blood flow to the brain. Several studies have demonstrated a relationship between hyperchloremia and death or disability observed in neurological diseases particularly ischemic stroke and ICH. The association between hyperchloremia and death or disability in patients with ischemic stroke and ICH is independent from the effect of patients' age or stroke severity. Hyperchloremia is also associated with occurrence of Acute Kidney injury in patients with subarachnoid hemorrhage and AKI was associated with higher mortality.

Hyperchloremia may induce metabolic acidosis which can results in intra- and extra- cellular acidosis in the brain leading to cytotoxicity via activation of enzymes and alteration in ionic movements and dysfunction of aquaporin-4 receptor leading to edema formation (9) and neural excitotoxicity.

Hyperchloremia may also augment pro-inflammatory response and modification of neutrophil and myeloperoxidase activity. Therefore, avoidance of hyperchloremia may be a therapeutic target in reducing death or disability among patients with ischemic stroke or ICH. The most effective strategy for reducing hyperchloremia is to reduce the chloride load through IV fluids.

A pilot study is proposed to identify the best" dose (ratio) of sodium chloride (0.9%) and sodium acetate (0.9%) mixture for reduction of hyperchloremia by using chloride efficient fluids in patients with acute stroke initiated within 12 hours of symptom onset and continued for 72hours.

Ethical and Regulatory Compliance:

This study will be conducted in accordance with all regulatory requirements. The trial will be conducted in compliance with the latest version of the Declaration of Helsinki, GCP, ICH and Ethics Review Committee guidelines and standards. Informed Consent Form will be administered in English and Urdu languages. A signed copy of the ICF will be provided to the subject for reference and record. Ethics Committee of Aga Khan Contact Person: Secretary ERC Research office Clinical Data Relevant Clinical Trial data will be transcribed from patient hospital file into study Case Report Forms (CRFs). Successively, all CRFs will be entered into Electronic Data Capture (EDC) software. All data collection, transmission and storage processes will be GCP compliant. Clinical data will be archived for 25 years after completion of study. Data access will be controlled by Principal Investigator and will only be granted to trained and delegated study staff.

Hypothesis:

Hyper chloremia is associated with poor outcome in Intracerebral Hemorrhage (ICT). Hyperchloremia is defined as serum chloride level of 110mmol/L or greater. This clinical study is assuming that, by increasing the ratio of Sodium-acetate to Sodium-chloride solutions in IV treatment, the incidence of Hyperchloremia can be lowered significantly. This result can be demonstrated by measuring serum chloride levels at Baseline, 24Hr, 48Hr and 72 Hours' time intervals and compare them between the three treatment and one Control arm.

Intervention (drug/biologic/device/behavioral):

Phase 2-dose finding Patients will be enrolled in the study and randomized into one of the four study treatment arms(target fluid administration rate 1 ml/kg/hour) initiated within 12 hours. IVF will be prepared in the main hospital pharmacy.

1. Sodium chloride (0.9%) referred as 0.9% NaCl for 72 hours post symptom onset (60-72 hourspost randomization);
2. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 3:1 ratio for 72 hours post symptom onset (60-72 hours post randomization);
3. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 2:1 ratio for 72 hours post symptom onset (60-72 hours post randomization);
4. Sodium chloride (0.9%) and sodium acetate (0.9%) mixture 1:1 ratio for 72 hours post symptom onset (60-72 hours post randomization).

   Primary Objective:

   To Determine the best dose of sodium chloride and sodium acetate mixture using efficient statistical strategy and its effects on outcome

   Primary Outcome:

   Persistent hyperchloremia:

   A complete chemistry panel will be performed at baseline, 24 hours, 48 hours, and 72 hours. "Persistent hyperchloremia within 72 hours will be the primary outcome. Patients with an increased serum chloride at either baseline, or 24, 48, or 72 hours after randomization were identified. Hyperchloremia will be defined by serum chloride of 110 mmol/L or greater consistent with previous studies.1-5 We will further grade hyperchloremia into one occurrence or two or more occurrences within first 72 hours as "persistent hyperchloremia". investigators anticipate that rate of persistent hyperchloremia will be 10-15% based on ATACH 2 and ALIAS 1 and 2 studies in patients with intracerebral hemorrhage and ischemic stroke, respectively.

   Acute Kidney Injury:

   investigators will ascertain and grade AKI severity after randomization based on the guidelines provided by the acute kidney injury network (AKIN) classification.8,9 Severity of AKI will be based on increase in serum creatinine levels from baseline and Urine Output. stage 1; ≥ 0.3 mg/dL (≥26.4 µmol/l) or A percentage increase in serum creatinine of 50% or greater (1.5 - 2-fold increase from baseline) stage 2; > 2 to 3-fold increase, stage 3; > 3-fold increase in serum creatinine. Or Oliguria: Urine output < 0.5 mL/kg per hour) for > 6hrs

   Secondary Outcome/Objectives:

   The secondary end point will be the mean score for disability on the utility-weighted modified rankin score (UW-mRS) at 90 days. UW-mRS weights the mRS against a health utility scale that reflects the spectrum between perfect health (a score of 1) and outcomes worse than death (where death isa score of 0 and negative values indicate an outcome worse than death).10,11 Thus, the UW-mRS ranges from 0 (death) to 10 (no symptoms or disability) and indicates the value to patients, families, and health providers of the long-term disability outcome, across a broad range from fully normal, through varying degrees of disability, to death.

   Additional secondary endpoints include:

   Metabolic alkalosis: Metabolic alkalosis will be defined by arterial pH >7.45 and HCO3- is >28 mmol/l.12,13

   All Serious Adverse Events:

   An Adverse Event is serious IF it leads to death or serious deterioration in the health of a subject that resulted in a life-threatening illness or injury, permanent impairment of a body structure or a body function, hospitalization or prolongation of existing hospitalization, medical or surgical intervention to prevent permanent impairment to a body structure or a body function and/or caused congenital anomaly or birth defect. All SAEs will be reported to the Sponsor, ERC, Hospital Incident Reporting system (AEMS) within 24 Hours of Investigator awareness and Regulatory body NIH/NBC/DRAP as soon as possible.
   * Ethics Committee can suspend/discontinue study if greater than acceptable risk is posed to the safety of participants.
   * Regulatory Authorities can also suspend/terminate study progress.
   * Sponsor may discontinue the study at any time with prior written notification.

   Risks and Side Effects:

   There are risks to taking part in any research study. There may also be other problems (also called side effects) we do not know about yet. If we learn about new important risks and side effects, we will inform the subject including any new information that may affect subject's decision to continue taking part in the study.

   Subjects may undergo a catheter-based procedure to remove the clot from the blood vessel (regardless of study participation).
   * There is a risk that any of the IV fluids will increase the fluid in subject's lungs which may require medication called diuretics to remove the fluids from lungs.
   * There is a risk that any of the IV fluids will make the kidney function worse which may require changing the IV fluids and additional treatment as considered appropriate by the doctor.
   * There is a risk that any of the IV fluids will cause increased acidity or alkalinity of the blood which may require discontinuation of the IV fluids and additional treatment as considered appropriate by the doctor.
   * There can be infection at the injection site, a dislodged IV catheter, or a collapsed vein when receiving any IV fluids. All of these are easily corrected or treated.
   * Finally, the experimental interventions in this study may have side effects that no one knows about yet.

   Settings:

   ALL clinical trial related interactions and investigations will be conducted in Aga Khan Hospital only.

   Relevant departments include Emergency Department, Neurology Department, Wards,Stroke Units, Main Lab and Out-Patient Clinics.

   Randomization and Elimination of Bias:

   A stratified randomization will be performed based on initial diagnosis of ischemic stroke or intracerebral hemorrhage. Patients will be randomized in permuted blocks of size 4 matched byclinical site (quadruplets) to 0.9% NaCl or one of the three doses of 0.9% NaCl: Na-acetate. Although patients were also randomized concurrently to 0.9% NaCl to preserve the blinding and to eliminate other possible temporal biases, only the 0.9% NaCl: Na-acetate arms will be involved in the section procedure. Furthermore, outcome assessments such as AE/SAE, degree of disability and MRS score will be performed by blinded and Independent medical staff to eliminate bias.
   * Total Sample size is 80 subjects (20 subjects per treatment arm)
   * Enrolment duration is 1year
   * Follow-Up duration is 3 months for each subject
   * Total study duration will be 18 months.

   Statistical assumptions:

   The dose finding trial will have Response Adaptive Randomization (RAR) updated beginning at 50 subjects enrolled and updated every 25 subsequent enrollments to a maximum sample size of 72 patients. The randomization will be after stratification based on ischemic stroke and intracerebral hemorrhage. The currently proposed design was selected because it collects information across a range of treatments, randomizes an increasing number of patients to the "best" arm in proportion to the amount of information available about the different treatments and quantifies the likelihood of success should a Phase III study be initiated. The chosen approach is expected to control for type 1 error at 10% and allows for greater than 80% power in all conditions tested.

   Statistical analysis:

   investigators will compare various measures of hyperchloremia between the four groups. Hyperchloremia will be defined by serum chloride ≥110 mmol/L at either baseline, or 24, 48, or 72 hours after randomization consistent with existing literature and into 1 occurrence or ≥2 occurrences within first 72 hours. Metabolic acidosis (serum bicarbonate of < 22 mmol/L consistent with previous studies) will also identified at same timepoints after randomization. investigators will also calculate area under the curve (AUC) to provide a summary of serum chloride levels over the 72-hour period.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Onset of new neurological deficits within 24 hours

NIHSS score of 4 or more

GCS score of 5 or more

CT scan demonstrates intraparenchymal hematoma with manual hematoma volume measurement <60 cm3 OR CT scan consistent with Ischemic Stroke

Exclusion Criteria:

received Intravenous fluids for greater than 8 hours

Baseline Serum Chloride is greater than 110 mmol/L

Acute Kidney Injury

History of Chronic Renal Failure

Requirement of Hemodialysis or Peritoneal Dialyses Prior to Randomization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
hyperchloremia into one occurrence or two or more occurrences within first 72 hours hyperchloremia" | 72 hours
  hyperchloremia into one occurrence or two or more occurrences within first 72 hours hyperchloremia"

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD WASAY, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
will share data after study completion